CLINICAL TRIAL: NCT07162025
Title: Development of a Specific Infant Formula for Babies Born by Caesarean Section
Brief Title: Improving Nutrition for Babies Born by Caesarean Section
Acronym: SPECIFI-C
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00676-43
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Breastfeeding Mothers of Legal Age; Their Babies Under 6 Months Old Born Vaginally
Keywords: caesarean section; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples and human breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ambition of the project is to help with the primal colonisation of babies born by caesarean section and to improve the lipid composition of an infant formula, in order to reduce the short- and long-term health problems associated with caesarean births. This population, which represents around 20% of babies born in France, has not yet received any specific care to date.

The study aims to develop an optimized infant formula. It includes: (1) isolation of probiotics from breast milk from nursing mothers and stool samples from their babies born vaginally, (2) formulation of an improved milk enriched with physiological lipids and selected probiotics, and (3) preclinical evaluation of its beneficial effects in a cesarean birth model.

DETAILED DESCRIPTION:
The perinatal period represents a critical window during which the establishment of the infant gut microbiota plays a central role in host physiology and immune system development. Cesarean delivery is associated with altered vertical transmission of maternal microbiota, leading to dysregulated host-microbiota interactions and impaired homeostasis. Epidemiological evidence indicates that disturbances in early-life colonization are linked to an increased risk of developing various non-communicable diseases later in life.

Modern obstetric practices, while highly effective in reducing birth complications, have resulted in a high prevalence of cesarean deliveries. Several strategies have been explored to restore the microbiota of cesarean-born infants, including maternal vaginal or fecal microbiota transfer, but these approaches raise significant safety concerns. Breastfeeding has been shown to partially restore the gut microbiota of cesarean-born infants; however, breastfeeding rates are lower after cesarean section than after vaginal delivery, largely due to postnatal complications that interfere with breastfeeding initiation. Although specific infant formulas already exist for certain populations, none are currently designed to address the impaired primary colonization observed in cesarean-born infants.

The SPECIFI-C project has been designed to fill this gap by developing an innovative infant formula tailored to the specific needs of this population. The strategy focuses on two main components: (i) optimization of the microbiological fraction through supplementation with beneficial microorganisms isolated from human breast milk and infant feces, and (ii) optimization of the lipid fraction by incorporating bioactive lipids such as docosahexaenoic acid (DHA) and alkylglycerols, which are naturally present in breast milk but absent from current formulas.

The ultimate objective is to provide a safe and effective nutritional intervention that promotes healthy gut colonization and supports immune and physiological development in cesarean-born infants. By targeting a population that represents approximately 20% of births in France, the project aims to contribute to more precise and personalized nutrition strategies, with the potential to reduce both short- and long-term health risks associated with cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding mothers:

Aged 18 years and older Breastfeeding for less than 6 months Not having taken probiotics in the 6 months prior to sampling Not having taken antibiotics in the 6 months prior to sampling No chronic medical conditions Not undergoing chronic treatment No history of gestational diabetes Body mass index (BMI) below 25 at the start of pregnancy Having given their consent to participate in the study and to the collection of their baby's stool samples Not deprived of liberty or placed under guardianship

- Babies: Aged less than 6 months Born vaginally Born at term or at least 37 weeks of pregnancy Exclusively breastfed Not having received intrapartum antibiotic treatment Having no known medical conditions Not receiving any medical supplements other than conventional vitamins Whose mothers meet the inclusion criteria detailed above

Exclusion Criteria:

Breastfeeding mothers:

* Under the age of 18
* Breastfeeding for 6 months or more
* Having been on antibiotic therapy in the 6 months prior to sampling
* Having taken probiotics in the 6 months prior to sampling
* Having a chronic illness
* Undergoing chronic treatment
* Who have developed gestational diabetes
* Who have a BMI greater than 25 at the start of pregnancy
* Who have given their consent to participate in the study (breast milk collection) but not to the collection of their baby's stool samples
* Who are deprived of their liberty or under guardianship.

Babies:

* Aged over 6 months
* Born by caesarean section
* Born before 37 weeks of pregnancy
* Not exclusively breastfed
* Having undergone intrapartum antibiotic treatment
* Taking medical supplements other than conventional vitamins
* Presenting with any type of pathology
* Whose mothers meet the non-inclusion criteria detailed above
* Receiving medical supplementation other than conventional vitamins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breastfeeding mothers and their babies under 6 months old
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of the viability of supplemented probiotic microorganisms (CFU/g) and levels of bioactive lipids in the experimental infant formula specifically designed for cesarean-born infants | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- INRAE, Jouy-en-Josas, France

IPD SHARING:
Plan to Share IPD: No